CLINICAL TRIAL: NCT01613339
Title: Body Awareness Therapy for People With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro County Council (Other Government)
Collaborators: Norrbacka-Eugenia Foundation (Other)
Responsible Party: Principal Investigator, Anette Forsberg, PhD, Researcher, RPT, Örebro County Council
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AF-1-2011
Record Dates: First submitted 2012-04-16; First posted 2012-06-07 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-05

CONDITIONS: Stroke
Keywords: stroke; postural control; body awareness therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Body awareness therapy (Experimental)
  Interventions: Other: Balance training using Body awareness therapy
- Control (No Intervention)

INTERVENTIONS:
Other: Balance training using Body awareness therapy — Once a week, 1 hour for 8 weeks.Body awareness training may be performed by physiotherapist. Exercises are performed in standing, sitting and lying. Example of exercises are weight-balancing in standing and relaxation exercises.
  Arms: Body awareness therapy

SUMMARY:
Affected balance capacity is common after a stroke due to paresis and sensory disturbances. The affected balance capacity may cause walking disturbances, falls and decreased mobility. Balance may be improved by physical therapy. A possible method for balance training is body awareness therapy, that was introduced in Sweden by Jacques Dropsy and Gertrud Roxendal. Earlier body awareness therapy was mostly used in psychiatric care but in the recent years the method has been used for people with long-tern pain, amputations and multiple sclerosis. Body awareness therapy includes exercises in lying, sitting and standing. Focus of the exercises are awareness of one´s movement behaviour, breathing patterns, resources and limitations. Postural control is an essential part in the exercises. Body awareness therapy could be used for people with stroke as a way to improve postural control. The aim of this study is to investigate if balance training using body awareness therapy can improve balance and walking in people after stroke. The interventions consists of body awareness therapy once a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed stroke more than 6 months ago. Walking capacity of 100 meter with or without assistive device.

Exclusion Criteria:

* Medical or cognitive impairment that prohibits participating in the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mialinn Arvidsson Lindvall, RPT, MSc, Principal Investigator — Family Medicine Research Centre, Örebro county council; Anette Forsberg, PhD, Study Chair — Family Medicine Research Centre, Örebro county council
Locations (1):
- Primary Health Care Centres, Örebro, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data collection was performed in the following order due to practical reason at four primary health care centres in Örebro county council; Kumla Primary health care center, October 2011- January 2012, Karla Primary health care centre, March 2012-June 2012, Nora and Brickegården Primary health care centre September 2012 to December 2012.
Groups:
- Body Awareness Therapy: Balance training using Body awareness therapy : Once a week, 1 hour for 8 weeks.Body awareness training may be performed by physiotherapist. Exercises are performed in standing, sitting and lying. Exemple of exercies are weight-balancing in standing and relaxation exercises.
- Control: No specific treatment.
Period: Overall Study
Arm/Group | Body Awareness Therapy | Control
Started | 24 | 22
Completed | 21 | 21
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Body Awareness Therapy | Control | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 10 | 24
  >=65 years | 10 | 12 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (11) | 66 (9) | 64 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 12 | 15 | 27
Region of Enrollment [Number; unit: participants]
  Sweden | 24 | 22 | 46

OUTCOME MEASURES:

1. Secondary Outcome: Timed Up and Go Test
Description: test of functional mobility. Time is taken in seconds. The participants sits on a chair with armrests are then asked to rise, walk 3 meters, turn and walk back and sit down.
Time Frame: Change from baseline in Timed Up and Go test at 9 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Body Awareness Therapy | Control
Number analyzed (Participants) | 21 | 21
seconds | 13.7 (7.3) | 17.6 (9.1)

2. Primary Outcome: Bergs Balance Scale
Description: Test of functional balance. Includes 14 items all graded 0-4 where 0 indicate larger impairment. Total score is used here, maximum 56 and minimum 0.
  The Berg balance scale was developed for older patients but is a much used meausure of dynamic and static functional balance.
Time Frame: Change from baseline in Bergs balance scale at 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Body Awareness Therapy | Control
Number analyzed (Participants) | 21 | 21
units on a scale | 52.3 (4.8) | 47.8 (7.4)

3. Secondary Outcome: Activities-specific Balance Confidence Scale
Description: 16 item questionnaire that investigates balance self-efficacy. Each items is a question; How secure are you that you will not fall when you...sweep the floor? The participant are asked to grade his/hers feeling of secutiry from 0, 10, 20 and so on up to 100. 0 is regarded low balance self-efficacy. The item responses are summed and divided by 16.
Time Frame: Change from baseline in Activities-specific Balance confidence scale at 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Body Awareness Therapy | Control
Number analyzed (Participants) | 21 | 22
units on a scale | 68.6 (20.3) | 59.1 (22.0)

ADVERSE EVENTS:
Groups:
- Body Awareness Therapy, Control: group training. Controls were asked to continue with their lifestyle.
Arm/Group | Body Awareness Therapy, Control
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No